CLINICAL TRIAL: NCT01992354
Title: Development of an Integrated PET/MR System, Accessories and Components
Brief Title: Development of an Integrated Positron Emission Tomography/Magnetic Resonance (PET/MR) System, Accessories and Components
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114-2013-GES-0012
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Indication for a PET CT Exam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): Evaluation of PET MR device for image assessment and device performance
  Interventions: Device: PET MR Device

INTERVENTIONS:
Device: PET MR Device — GE PET/MRI system

SUMMARY:
The PET/MR device components and accessories are under development in order to optimize, validate and improve the design including improving the quality of images. The purpose of this study is:

* Aim 1: Perform iterative evaluations of the device (including features and components) to optimize device performance and assess feasibility of new features;
* Aim 2: Perform activities in support of design validation as needed for regulatory submission;
* Aim 3: Evaluate device complaints and analyze potential causes.

DETAILED DESCRIPTION:
This is a non-randomized, non-statistically powered, single-site, prospective study designed to gather imaging data for design optimization, regulatory submission and future product development of an investigational hybrid PET/MRI scanner. Subjects will undergo a clinically indicated PET/CT exam subsequent to tracer administration. Once clinical imaging is complete, subjects will be transported to the PET/MR scanner at the General Electric (GE) Facility for additional imaging. No additional pharmaceuticals or ionizing radiation will be utilized as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a clinical indication for a PET/CT exam
* Subject must be at least eighteen (18) years of age; and
* Subject must be able to hear and understand instructions without assistive devices; and
* Subjects must be ambulatory, and able to walk 350 feet without any assistive devices and climb 2 steps; and
* Subject must be able to provide identification with photograph; and
* Female subjects with negative urine pregnancy test performed within 24 hours prior to the clinical PET/CT imaging; and
* Subject must provide written informed consent; and
* Subject has the necessary mental capacity to understand instructions, and is able to comply with protocol requirements; and
* Subject is able to remain still for duration of imaging procedure (approximately 60 minutes total for PET/MRI); and
* Subject must be able to participate in a PET/MR imaging session within 1 hour of concluding their PET/CT exam

Exclusion Criteria:

* General Electric Healthcare (GEHC) employees; or
* GEHC contractors; or
* Healthcare providers (Any person in a position to purchase, lease, recommend, use, prescribe or arrange for the purchase or lease of any GEHC product or service that is reimbursable under any government program or private health insurance) or employees/contractors of medical device companies (as determined by self-report); or
* Female subjects with known or suspected pregnancy; or
* Subjects who have any axial diameter larger than 55 cm; or
* Subjects with a weight greater than 227 kgs; or
* Subjects who currently have, or have ever had a Cardiac Pacemaker or Defibrillator with implanted components; or
* Subjects who are currently undergoing a gastrointestinal study involving swallowing of camera pill or similar device; or
* Subjects who have any of the conditions below at the time of the scan session:

  * Prior negative experience or problem related to a previous MRI examination
  * Eye injury involving a metallic object
  * Potential for metal to be in body due to a previous injury involving metallic objects
  * Taking fertility medication or having fertility treatment
  * Cochlear, otologic or other ear implant
  * Insulin or other infusion pump
  * Implanted drug infusion device
  * Any type of prosthesis (eye, penile, etc)
  * Swan-Ganz or thermodilution catheter
  * Any metallic fragment or foreign body
  * Artificial or prosthetic limb
  * Bone/joint pin, screw, nail, wire, plate, etc
  * Neurostimulation system
  * Surgical staples, clips, or metallic sutures;
  * Implanted cardioverter defibrillator (ICD);
  * Magnetically activated implant or device;
  * Vascular access port and/or catheter;
  * Medication patch (Nicotine, Nitroglycerine);
  * Internal electrodes or wires;
  * External electronic medical device
  * Bone growth/bone fusion stimulator
  * Radiation seeds or implants
  * Heart valve prosthesis
  * Spinal cord stimulator
  * Eyelid spring or wire
  * Wire mesh implant
  * Tissue expander (e.g. breast)
  * Aneurysm clip(s)
  * Joint replacement (hip, knee, etc…)
  * Vascular or other stent(s), filter(s) or coil(s)
  * Intra-uterine device, diaphragm or pessary
  * Shunt (spinal or intraventricular)
  * Loose dental fillings
  * Dental fillings or crowns placed in the past 30 days
  * Tattoo or permanent makeup
  * Any implant
  * Breathing problem or motion disorder
  * Claustrophobia or panic attacks
  * Hearing Aid
  * Body piercing jewelry
  * Dentures or partial plates
  * External medical hardware (e.g. orthopedic braces)
  * Orthodontic appliances (e.g. braces, expanders)
  * Known or past allergic reactions to latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Prost, PhD, Principal Investigator — Froedtert Hospital
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PET/MR System: Evaluation of Positron Emission Tomography/Magnetic Resonance (PET/MR) device for image assessment and device performance
  PET MR Device: General Electric (GE) PET/MRI system
Period: Overall Study
Arm/Group | PET/MR System
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: PET/MR Scan Obtained
Description: One PET/MR scan per subject should be obtained. The scan images are evaluated by a subject matter expert for adequate diagnostic quality.
Time Frame: One (1) day
Measure: Number; unit: scans completed
Groups:
- PET/MR System: Evaluation of PET MR device for image assessment and device performance
  PET MR Device: GE PET/MRI system
Arm/Group | PET/MR System
Number analyzed (Participants) | 4
scans completed
  Scans supporting Aim 1 | 5
  Scans supporting Aim 2 | 0
  Scans supporting Aim 3 | 0

2. Secondary Outcome: Device Complaints
Description: Number of device complaints reported during a scan
Time Frame: One day
Measure: Number; unit: Device complatints reported
Arm/Group | PET/MR System
Number analyzed (Participants) | 4
Device complatints reported | 0

ADVERSE EVENTS:
Time Frame: One (1) day
Description: One (1) day, during diagnostic procedure
Arm/Group | PET/MR System
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No